CLINICAL TRIAL: NCT04492059
Title: Use of Blood Flow Restriction Therapy in Perioperative Rehabilitation Following Achilles Tendon Rupture
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No patients
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Erickson Andrews, M.D., Principal Investigator, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BFR Achilles Tendon
Record Dates: First submitted 2020-06-07; First posted 2020-07-30 (Actual); Last update posted 2023-02-02 (Actual); Status verified 2023-01

CONDITIONS: Achilles Tendon Rupture; Achilles Tendon Surgery
Keywords: Blood flow restriction; physical therapy; Achilles tendon; Achilles tendon rupture; Achilles tendon repair
MeSH Terms: interventions — Physical Therapy Modalities

STUDY DESIGN:
Intervention Model Description: Patients will be assigned to the blood flow restriction augmented physical therapy group following surgery or will undergo the usual physical therapy. Various measurements will be taken at follow up appointments as well as patient reported outcomes and compared between the two groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Blood flow restriction augmented physical therapy (Experimental): The group will undergo traditional physical therapy with the augment of blood flow restriction therapy under the supervision of trained physical therapists.
  Interventions: Device: Blood flow restriction augmented physical therapy
- Traditional physical therapy (Active Comparator): The group will undergo traditional physical therapy without the augment of blood flow restriction therapy under the supervision of trained physical therapists.
  Interventions: Other: Physical therapy

INTERVENTIONS:
Device: Blood flow restriction augmented physical therapy — Using a blood flow restriction cuff during physical therapy. It is a pressurized cuff that is used to decrease the amount of oxygen that is available to the muscle during exercise. This stimulates the muscle to believe it is in an anoxic state and can produce greater strength and hypertrophy with fewer reps and less weight which would mean less stress on a surgically repaired tendon.
  Arms: Blood flow restriction augmented physical therapy
Other: Physical therapy — Completing traditional physical therapy.
  Arms: Traditional physical therapy

SUMMARY:
The purpose of this study is to examine the effect of utilizing blood flow restriction (BFR) therapy in the rehabilitation of Achilles tendon rupture (ATR). Muscle atrophy occurs following Achilles tendon rupture, whether managed non operatively or operatively, which has implications on patient outcomes. The goal of physical therapy in the perioperative period is to regain and ultimately return to activity. BFR has been proposed to reduce atrophy and maintain strength, which would theoretically mitigate the deconditioning effects of an injury on surrounding musculature. BFR is proposed to work by restricting arterial inflow leading to an oxygen depleted environment and the ability to induce muscle adaption at lower maximum repetition via reactive hyperemia and induction of growth cytokines, thus leading to muscle hypertrophy.

The goal of this investigation is to determine if using BFR as an adjunct in physical therapy following ATR would reduce muscular atrophy and lead to increased and expedited strength gains. Additionally, the investigators would like to determine if BFR accelerates the rehabilitation process and allows patients to perform standard rehabilitative functional tests and return to play sooner. Furthermore, the investigators will investigate patient reported outcomes metrics.

The investigators hypothesize that the BFR group will have significantly greater strength gains at all time points in both non operatively and operatively treated ATR. Previous studies have shown that BFR has potential in increasing Achilles tendon stiffness, tendon cross-sectional area, muscle strength and muscle hypertrophy. However, there is a lack of evidence regarding the use of BFR in both the pre and postoperative period specifically relating to ATR. The investigators believe that the use of BFR in the perioperative period surrounding an Achilles tendon rupture and ATR has the potential to significantly decreased muscle atrophy, improve patient satisfaction and lead to earlier return to sport.

DETAILED DESCRIPTION:
Following diagnosis of ATR, attending surgeons will discuss treatment options with the patient and determine their course of treatment to be operative or non-operative. Patients will then be randomized via computer to prospectively undergo ATR rehabilitation using conventional therapy or conventional therapy with a BFR adjunct by physical therapists already trained in BFR with extensive experience in ATR rehabilitation. There will be no incentive provided for participation by the therapists and the therapists may opt out of using BFR at any point. Treatment groups will undergo similar protocols with the only difference being the use of BFR as an adjunct to their rehabilitation. The protocol for using the BFR cuff will be similar to previous studies examining BFR in lower extremity injuries, with adaptation to the postoperative protocol specific to the Achilles tendon. More specifically the physical therapists will be provided with a tourniquet that includes a pressure monitor. The skin will be protected with a sleeve and the cuff will be placed in the thigh well proximal to the knee joint. The investigators will begin by determining the patient's limb occlusion pressure, which is conducted automatically by the cuff via built in doppler. Once this is done the cuff will be inflated to 80% of the limb occlusion pressure, which is the currently accepted recommendation in the literature and sufficient to achieve the desired effect of blood flow restriction.

For non-operative candidates the investigators will begin their rehabilitation and physical therapy immediately following their initial office visit. Participants will have follow-up appointments at two-weeks, six-weeks, three-months and six-months. During these follow-up appointments the investigators will assess calf strength, calf circumference, ankle range of motion, current pain and function level. Additionally, the investigators will conduct testing at the end of the therapy sessions to ensure patients are prepared to return to sports.

For operative candidates the investigators will schedule their surgery at the earliest convenience and availability following their initial office visit. Participants will begin their rehabilitation and physical therapy immediately following their surgery. Participants will have follow-up appointments at two-weeks, six-weeks, three-months and six-months. During these follow-up appointments the investigators will assess calf strength, calf circumference, ankle range of motion, current pain and function level. Additionally, the investigators will conduct testing at the end of the therapy sessions to ensure patients are prepared to return to sports.

In both operative and non-operative rehabilitation, therapy will consist of a structured program progressing from range of motion to strength training and then functional tests. Both those randomized to conventional therapy and those randomized to conventional therapy with BFR adjunct will follow the same protocol with the only variable being the use of BFR. Again, the BFR group will have the cuff inflated per protocol outlined above, this will be under the guidance of trained physical therapists.

Throughout this protocol patient will have their initial/pre-operative visit to establish care and set up surgery and follow-up appointments at two-weeks, six-weeks, three-months and six-months. All data collection and testing during these follow-up appointments will be obtained with a handheld device and will add less than five minutes to clinic visits.

ELIGIBILITY:
Inclusion Criteria:

* patients aged 18-65 who suffered an achilles tendon rupture.
* Patients with achilles tendon rupture that are being treated operatively and non-operatively.

Exclusion Criteria:

* undergoing a revision procedure
* other concomitant injuries of the same leg
* have a history of deep vein thrombosis
* peripheral vascular disease
* neurovascular injury to the extremity
* are unable to tolerate BFR treatment
* have a leg circumference greater than the largest available tourniquet circumference of 96.52 cm
* unable to complete physical therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-03-25 (Actual); Study Completion 2022-03-25 (Actual)

PRIMARY OUTCOMES:
Change in plantarflexion strength from baseline | Measured at six-week, three-month and six-month postoperative visits
  Plantarflexion strength to be measured via dynamometer

SECONDARY OUTCOMES:
Change in range of motion | Measured at six-week, three-month and six-month postoperative visits
  Dorsiflexion and plantar flexion measured with goniometer
Achilles Tendon Total Rupture Score | Measured at initial visit, six-week, three-month and six-month postoperative visits
  Score used to assess disability and function of patients with achilles tendon rupture. Range is 0-100, with 100 being full function and no deficits.
Pain on the visual analog score | Measured at initial visit, six-week, three-month and six-month postoperative visits
  Patient self assessment of current pain. Range is 0 - 10, with 0 being no pain and 10 being the worst pain the patient has experienced.
PROMIS pain scores | Measured at initial visit, six-week, three-month and six-month postoperative visits
  Patient reported outcomes using the PROMIS algorithm. 50 is average, the standard deviation is 10. Range is 0-100. A score of 60 would indicate one standard deviation more pain than average.
PROMIS function scores | Measured at initial visit, six-week, three-month and six-month postoperative visits
  Patient reported outcomes using the PROMIS algorithm. 50 is average, the standard deviation is 10. Range is 0-100. A score of 60 would indicate one standard deviation better function than the average.
PROMIS depression scores | Measured at initial visit, six-week, three-month and six-month postoperative visits
  Patient reported outcomes using the PROMIS algorithm. 50 is average, standard deviation is 10. Range is 0-100. A score of 60 would indicated one standard deviation more depression than average.
Change in calf circumference | Measured at initial visit, six-week, three-month and six-month postoperative visits
  Circumference measurements of the calf

CONTACTS AND LOCATIONS:
Overall Officials: Erickson Andrews, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Hospital, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Heikkinen J, Lantto I, Flinkkila T, Siira P, Laine V, Niinimaki J, Ohtonen P, Leppilahti J.
- [Background] Wernbom M, Augustsson J, Raastad T. Ischemic strength training: a low-load alternative to heavy resistance exercise? Scand J Med Sci Sports. 2008 Aug;18(4):401-16. doi: 10.1111/j.1600-0838.2008.00788.x. Epub 2008 May 3. PMID 18466185
- [Background] Centner C, Lauber B, Seynnes OR, Jerger S, Sohnius T, Gollhofer A, Konig D. Low-load blood flow restriction training induces similar morphological and mechanical Achilles tendon adaptations compared with high-load resistance training. J Appl Physiol (1985). 2019 Dec 1;127(6):1660-1667. doi: 10.1152/japplphysiol.00602.2019. Epub 2019 Nov 14. PMID 31725362
- [Background] Yow BG, Tennent DJ, Dowd TC, Loenneke JP, Owens JG. Blood Flow Restriction Training After Achilles Tendon Rupture. J Foot Ankle Surg. 2018 May-Jun;57(3):635-638. doi: 10.1053/j.jfas.2017.11.008. Epub 2018 Feb 21. PMID 29477554
- [Background] Ladlow P, Coppack RJ, Dharm-Datta S, Conway D, Sellon E, Patterson SD, Bennett AN. Low-Load Resistance Training With Blood Flow Restriction Improves Clinical Outcomes in Musculoskeletal Rehabilitation: A Single-Blind Randomized Controlled Trial. Front Physiol. 2018 Sep 10;9:1269. doi: 10.3389/fphys.2018.01269. eCollection 2018. PMID 30246795
- [Background] DePhillipo NN, Kennedy MI, Aman ZS, Bernhardson AS, O'Brien L, LaPrade RF. Blood Flow Restriction Therapy After Knee Surgery: Indications, Safety Considerations, and Postoperative Protocol. Arthrosc Tech. 2018 Sep 24;7(10):e1037-e1043. doi: 10.1016/j.eats.2018.06.010. eCollection 2018 Oct. PMID 30377584
- [Background] Noordin S, McEwen JA, Kragh JF Jr, Eisen A, Masri BA. Surgical tourniquets in orthopaedics. J Bone Joint Surg Am. 2009 Dec;91(12):2958-67. doi: 10.2106/JBJS.I.00634. PMID 19952261
- [Background] Clark BC, Manini TM, Hoffman RL, Williams PS, Guiler MK, Knutson MJ, McGlynn ML, Kushnick MR. Relative safety of 4 weeks of blood flow-restricted resistance exercise in young, healthy adults. Scand J Med Sci Sports. 2011 Oct;21(5):653-62. doi: 10.1111/j.1600-0838.2010.01100.x. Epub 2010 Mar 11. PMID 21917016
- [Background] Madarame H, Sasaki K, Ishii N. Endocrine responses to upper- and lower-limb resistance exercises with blood flow restriction. Acta Physiol Hung. 2010 Jun;97(2):192-200. doi: 10.1556/APhysiol.97.2010.2.5. PMID 20511128